CLINICAL TRIAL: NCT01025063
Title: Use of Spectral OCT in Combination Therapy
Acronym: Spectral OCT
Status: Completed | Type: Observational
Sponsor: Barnes Retina Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Rhonda Weeks, Gaurav K. Shah, MD, Barnes Retina Institute
Other Study IDs: CBPD952AUS18T
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Choroidal Neovascularization
Keywords: Spectral OCT; Choroidal Neovascularization; Lucentis; Visudyne; PDT; anti-VEGF
MeSH Terms: conditions — Choroidal Neovascularization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Lucentis (PRN group)
- Lucentis (3 Injections over three months)
- PDT (Reduced Fluence) and Lucentis

SUMMARY:
This study will investigate the safety and efficacy of treatment of choroidal neovascularization (CNV) due to age-related macular degeneration (AMD) with a combination of ranibizumab (Lucentis) and verteporfin PDT (Visudyne), as compared with ranibizumab monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Patients with visual acuity of 20/40-20/320 in the study eye
* Subfoveal choroidal neovascularization (CNV) must be at least 50% of the total lesion size.
* Total area of lesion components other that CNV must be less than 50% of the total lesion size.
* The lesion must be < 5400microns in greatest linear dimension (GLD).
* Lesion size < 10 DA
* Occult with no classic CNV lesions must have presumed recent disease progression:

  1. Blood associated with the lesion at baseline
  2. Loss of visual acuity in the previous 3 months: a: > 5 letter loss (ETDRS equivalent) or b: 2 or more lines using a snellen or equivalent chart
  3. > 10% increase in GLD as assessed by fluorescein angiography in the previous 3 months

Exclusion Criteria:

* Presence of angioid streaks, presumed ocular histoplasmosis syndrome, pathologic myopia (-8 or more with evidence of posterior segment abnormalities consistent with pathologic myopia), or CNV secondary to causes other than AMD
* Geographic atrophy in the study eye
* Tear (rip) of the retinal pigment epithelium
* Presence of fibrosis, hemorrhage, pigment epithelial detachments, or other hypofluorescent lesions obscuring greater than 50% of the CNV lesion
* Intraocular surgery within 6 weeks of enrollment
* Active or history of ocular inflammation or infection in the study eye within the last 30 days
* Subretinal hemorrhage > 50% of the total lesion
* History of submacular surgery, or transpupillary thermotherapy in the study eye
* Patients with intraocular pressure greater than 30 mm/Hg on 2 pressure-lowering medications
* Patients with severe disciform scarring
* History of intraocular surgery in the study eye including pars plana vitrectomy, except for uncomplicated cataract surgery within 60 days prior to screening
* History of YAG laser posterior capsulotomy in the study eye within 30 days prior to screening
* Inability to make study visits
* Advanced glaucoma, uncontrolled glaucoma in the study eye (defined as intraocular pressure, IOP ≥ 25 mmHg) despite treatment with two or more topical pharmacological anti-glaucomatous medication)
* Allergies to porphyrins or a known hypersensitivity to any component of Visudyne®
* Patients with porphyria
* Pregnancy or lactation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Barnes Retina Institute clinic
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
This pilot study observed anatomical measures which are currently not defined since the new technology is unclear in regards to what changes are seen at the level of the RPE and photoreceptors. | 3 months